CLINICAL TRIAL: NCT05223309
Title: Loose Thick Seton Suture Stimulate Rapid Healing and Lower Recurrence Rate in the Treatment of High Type Fistula in Ano
Brief Title: High Type Fistula in Ano, Use Staged Seton, Loose Thick Sutures
Status: Completed | Type: Observational
Sponsor: Jabir Ibn Hayyan Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Seton
Record Dates: First submitted 2021-10-19; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-05

CONDITIONS: Fistula in Ano
Keywords: High type; Seton; Loose thick sutures; Recurrance
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Usinf thick loose sutures in seton techingues — All patients were informed about doing fistulectomy and thick silk Seton suture placement for three months by excising the extrasphincteric part and putting the Seton suture to the intersphincteric part. Then, the second stage of operation includes the excision of the changing low type tract in which the silk Seton placed. We decrease the time of Seton placement in this study for three months to reduce the annoying symptoms of the patients. Therefore, the patient admitted to the operation theater after obtaining written consent. Most of the patients anesthetized by spinal anesthesia. In the operation theater, the patient assumed a lithotomy position
  . After that, the injection of a solution, which is a mixture of methylene blue dye and hydrogen peroxide into the external opening of the fistula, was done to find the internal opening. The exit of color dye or bubbles achieved to localized of inner opening from it after using intraoperative proctoscopy examination.

SUMMARY:
Fistula in ano is a chronic problem for the patients. It causes distressing because of foul odor and soiling with recurrent infection and discharge. Recurrence and anal sphincter injury were the most critical complications following surgery. Loose, thick Seton placement was the most promising surgical operation. To reduce the time of Seton placement, therefore, decreasing the suffering of patients from soiling and multiple dressing.

DETAILED DESCRIPTION:
Background: Fistula in ano is a chronic problem for the patients. It causes distressing because of foul odor and soiling with recurrent infection and discharge. Recurrence and anal sphincter injury were the most critical complications following surgery. Loose, thick Seton placement was the most promising surgical operation. To reduce the time of Seton placement, therefore, decreasing the suffering of patients from soiling and multiple dressing.

Patients and Methods: A retrospective study. One hundred patients with high type fistula in ano treated surgically in Al-Sader Medical city and Al-Najaf daily private clinic, Najaf city, Iraq from Feb 2018 to March 2019. Fistulography and magnetic resonance imaging have taken from all patients. After that, fistulectomy with loose, thick Seton suture placed for three months. Patients with the persistence of high fistula tract underwent a second surgery and third operation until complete healing.

ELIGIBILITY:
Inclusion Criteria:

* High type fistula in ano Recurrent high type fistula in ano Non abscess cases

Exclusion Criteria:

Low type fistula in ano below 16 years old

-

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Age distribution of patients showed that the highest rate of patients lies between the ages of 20-60 years adult population
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Rapid healing and less recurrent | 2 year
  usage of loose Seton in high type FIA

CONTACTS AND LOCATIONS:
Overall Officials: Samer Al-Hakkak, Ph.D., Study Chair — Jabir Ibn Hayyan Medical University
Locations (1):
- Samer Al-Hakkak, Najaf, An Najaf, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Share data
Time Frame: about 2 year
Access Criteria: document